CLINICAL TRIAL: NCT01450345
Title: Efficacy of Pre-operative Oral Pregabalin in Ambulatory Inguinal Hernia Repair for Post Operative Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Toh Charng Chee, Principle Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: toh2c79@Pregabalin
Record Dates: First submitted 2011-09-24; First posted 2011-10-12 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Inguinal Hernia; Postoperative Pain
Keywords: Clinical diagnosis of inguinal hernia; Patient undergo operation under daycare basis; ASA I-II; Written consent
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregabalin Group (Experimental): The patient under Group P will be serving with 150 mg of oral Pregabalin 1 to 2 hours prior to induction.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — The patient under Group P will be serving with 150 mg of oral Pregabalin 1 to 2 hours prior to induction.
  Other Names: Lyrica 150mg

SUMMARY:
The study carry out is to determine whether the use of oral pregabalin premedication to assess the analgesic efficacy, opiod sparing, adverse effect and clinical value in post-operative pain management.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of inguinal hernia
* Patient undergo operation under daycare basis
* ASA I-II
* Written consent

Exclusion Criteria:

* ASA > II
* Allergic reaction against gabapentin and/or pregabalin
* History of recurrent hernia repair.
* Patient who has taken analgesia prior to the surgery
* Liver failure
* Renal failure
* Pregnancy

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Study is constructed to determine whether the use of oral pregabalin premedication to assess the analgesic efficacy for post operative pain at Alert, 15, 30, 45, 60 and 120 min, Day 1, Day 2 and Day 3. | 3 days
  Efficacy: To compare the VAS score for pain after operation between the group at Alert, 15, 30, 45, 60 and 120 min, Day 1, Day 2 and Day 3.

SECONDARY OUTCOMES:
Opiod Sparing | 3 days
  Total amount of rescue medication requires
Side effect of medication | 3 days
  Severity of Post operative nausea and vomiting (PONV) graded with mild, moderare and severe(Vomiting) Side effect of medication includes headache, giddiness, visual disturbance, and difficulty in walking.

CONTACTS AND LOCATIONS:
Overall Officials: CharngChee Toh, MBBS, MRCS, Principal Investigator — University of Malaya
Locations (1):
- University Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia